CLINICAL TRIAL: NCT06919263
Title: Influencer E-Cigarette and Cannabis Marketing: a Survey-Based Experiment Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jennifer Unger, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: HS-19-00682-AM016; T33DT6620 (Other Grant/Funding Number: TRDRP)
Record Dates: First submitted 2025-03-20; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Electronic Nicotine Delivery Systems
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: Images featuring influencers promoting e-cigarettes alongside cannabis products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group (Active Comparator): Images featuring influencers promoting e-cigarettes alongside cannabis
  Interventions: Behavioral: Influencer marketing
- Placebo group (Active Comparator): Images featuring neutral profiles of influencers not using or displaying any substances
  Interventions: Behavioral: Influencer marketing
- Control (Active Comparator): Images featuring influencers promoting e-cigarettes alone
  Interventions: Behavioral: Influencer marketing

INTERVENTIONS:
Behavioral: Influencer marketing — Participants viewed survey-imbedded promotional images featuring influencers

SUMMARY:
Adolescent non-users of e-cigarettes and cannabis (N = 1,462) participated in the in-class survey-based experiment. They were randomly shown 3 pairs of images featuring influencers promoting e-cigarettes alongside cannabis, (experimental group), or no-substance use or display (placebo treatment), or e-cigarette promotion alone (control). After viewing each pair of images, participants rated perceptions of influencer credibility (i.e., honesty, trustworthiness, knowledge) on the scale of 0 (e.g., dishonest) to 100 (honest).

Susceptibility to use e-cigarettes was assessed after participants viewed all the images. These outcomes were then compared among participants who perceived influencers as credible and those who perceived influencers as non-credible.

DETAILED DESCRIPTION:
Adolescents (13-17 years of age) living in California were recruited by Tobacco Center of Regulatory Science at the University of Southern California (USC TCORS) to participate in the ADVANCE survey cohort focused on tobacco-related attitudes and behaviors. Participants completed the experiment, which was part of the survey at cohort's Wave 7, on Chromebooks in classroom. All participants provided informed consent and parental assent prior to participating in the experiment. The study was approved by the University of Southern California Institutional Review Board (HS-19-00682-AM016). Respondents were randomly shown 3 pairs of images featuring influencers promoting e-cigarettes (image 1) paired with cannabis (image 2), (experimental group), or no-substance use or display (two images featuring neutral profiles of influencers), (placebo treatment), or e-cigarette promotion (image 1) paired with a neutral profile (with no e-cigarette) of the influencer featured in image 1 (control).

ELIGIBILITY:
Inclusion Criteria:

* English fluency,
* Current California resident.

Exclusion Criteria:

Not meeting these criteria:

* English fluency,
* Current California resident.

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1462 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Perceptions of influencer credibility | assessed during the ~ 30-minute experiment, immediately after each of the three pairs of influencer images
  Perceptions of influencer credibility (i.e., honesty, trustworthiness, knowledge) were assessed using a 0 (e.g., dishonest) -100 (e.g., honest) scale that has been validated in prior research.
Susceptibility to use e-cigarettes | one-time assessment after the experimental exposure (immediately post-treatment)
  Susceptibility to use e-cigarettes was measured using the validated three-item scale adapted from Population Assessment of Tobacco and Health (PATH), and combined into one variable (α=0.93). Consistent with prior research, the measure was dichotomized with responses "definitely not" to all items being coded as "not susceptible" and responses "probably not," "probably yes", or "definitely yes" being coded as "susceptible."

CONTACTS AND LOCATIONS:
Overall Officials: Gina Klemm, Study Director — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States